CLINICAL TRIAL: NCT04924881
Title: Chinese Medicine for Residue Symptoms of COVID-19 Recovered Patients- A Double-blind, Randomized, Placebo-controlled Study
Brief Title: Chinese Medicine for Patients With LCOVID-19 Symptoms
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Lin Zhixiu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LCOVID study
Record Dates: First submitted 2021-06-10; First posted 2021-06-14 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Arm (Experimental): COVID Rehab Formula granules once daily for 8 weeks
  Interventions: Drug: COVID Rehab Formula granules
- Placebo Arm (Placebo Comparator): Placebo granules once daily for 8 weeks
  Interventions: Other: Placebo granules

INTERVENTIONS:
Drug: COVID Rehab Formula granules — COVID Rehab Formula granules once daily for 8 weeks
  Arms: Active Arm
Other: Placebo granules — Placebo granules once daily for 8 weeks
  Arms: Placebo Arm

SUMMARY:
COVID-19 has spread rapidly and now affects all over the world. On 11 March 2020, coronavirus disease 2019 (COVID-19) was declared a global pandemic by the World Health Organization (WHO).

Most of the infected people will develop mild to moderate illness, for example fever, cough, tiredness and joint pain etc. For some older people, and those with comorbidities like cardiovascular disease, diabetes, chronic respiratory disease, and malignancy are more likely to develop serious illness. Also long-term problems such as fatigue, breathlessness and joint pain experienced by survivors of COVID-19 after discharge from hospital.

Some clinical and pharmacological studies have suggested Traditional Chinese Medicine (TCM) has achieved remarkable therapeutic effect for active COVID cases of different severity during SARS epidemic in 2003. Also, some studies shown that using Chinese medicine interventions together with conventional treatment is more effective than using the conventional treatment alone in treating chronic fatigue syndrome.

Traditional Chinese Medicine (TCM) has a long history and played an important role in the prevention and treatment of several epidemic diseases. However, there is a lack of clinical study of using TCM to treat the residue symptom of COVID-19 recovered patients.

COVID-19 recovered patients will be screened and randomized into TCM group or placebo group for 8 weeks and followed by a post-treatment visits at week 12.

DETAILED DESCRIPTION:
Coronaviruses (CoV) are a large family of viruses that cause illness ranging from the common cold to more severe diseases. A novel coronavirus (nCoV) is a new strain that has not been previously identified in humans. COVID-19 has spread rapidly and now affects all over the world. As of 31 Jan 2021, over 100 million COVID-19 confirmed cases were reported worldwide, with more than 2 million related death.

Up to now, most frequently used therapies are corticosteroids, antiviral agents, antiviral/immunomodulatory drugs, serotherapy, anticoagulant and inflammation inhibitors. Recent studies reported that different kinds of residue symptoms were left after patient discharged from the hospital, such as fatigue, breathlessness and joint pain.

During SARS epidemic in 2003, the treatment of Traditional Chinese Medicine (TCM) has achieved remarkable therapeutic effect. Many different types of TCM have been proposed to treat COVID-19, of which the most famous are "three medicines and three formulae": Jinhua Qinggan Granule, Lianhua Qingwen Capsule/Granule, Xuebijing Injection; Lung Cleansing and Detoxifying Decoction, HuaShiBaiDu Formula and XuanFeiBaiDu Formula, which are mainly used for active COVID cases of different severity. Clinical and pharmacological studies have suggested their efficacy, safety and possible mechanisms in treating different stages of COVID-19, either used along with conventional treatment or independently.

For residual symptoms seen in COVID recovered patients, such as fatigue, dyspnoeaand insomnia, there are also studies suggesting that TCM may be helpful. Some studies shown that using Chinese medicine interventions together with conventional treatment is more effective than using the conventional treatment alone in treating chronic fatigue syndrome.

Liujunzhi Decoction (LJZD) and Shashen Maidong Decoction (SSMDD) are classic Chinese medicine formulae that have been used in China for hundreds of years. Their combination is proposed as the intervention of this trial because, from the perspective of Chinese medicine, the residual symptoms of COVID-19 can often be seen as the manifestation of "lung-spleen qi deficiency" or "qi and yin deficiency". ModifiedLJZD and SSMDD are the two most frequently recommended formulae versions in the recovery stage of COVID-19. This study is to evaluate the efficacy of using COVID Rehab Formula "CRF"(LJZD and SSMDD with variations) on the residue symptom of COVID-19 recovered subjects. To evaluate the efficacy of using COVID Rehab Formula "CRF" on the residue symptom of COVID-19 recovered subjects. COVID-19 recovered patients will be randomly assigned to TCM group or placebo group for study treatment 8 weeks and followed by a post-treatment visits at week 12.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 18;
* Have fatigue and one more residue symptoms (e.g. dyspnoea, sleep disturbance, cough, loose stool, abdominal distension, loss of appetite, dizziness, etc.) at least 5 weeks after discharge
* Patients are diagnosed with "lung-spleen qi deficiency"(肺脾氣虛) and/or"dual deficiency of qi and yin"(氣陰兩虛) by a Chinese Medicine Practitioner
* Voluntary written consent.

Exclusion Criteria:

* Still being SARS-CoV-2 positive
* Known severe medical conditions, such as cardiovascular, liver or renal dysfunction, diabetes mellitus, cancers, cerebrovascular diseases, blood system diseases;
* Impaired hematological profile and liver / renal function;
* No concomitant non-steroidal anti-inflammatory drugs (NSAIDs), steroids, antibiotics, prebiotics, probiotics within 4 weeks;
* Known allergic history to any Chinese herbal medicines;
* Known pregnancy or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The Change of Fatigue Severity Score | 8 weeks
  Improvement of residue COVID-19 symptoms of fatigue after study treatment at week 8, using a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. Scores range from 9 - 63; the higher the score, the greater fatigue severity.

SECONDARY OUTCOMES:
Long Term Symptom Assessment | 8 weeks
  Self-reported long term COVID-19 symptoms For the symptom questionnaire, participants will be asked to report newly occurring and persistent symptoms, or any symptoms worse than before COVID 19 development. The symptom assessment has 5 scale, from none to very severe.
The Change of Fatigue Severity Score (FSS) | 12 weeks
  FSS is a 9 item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. Scores range from 9-63; the higher the score, the greater fatigue severity.
Improvement of dyspnoea using modified British Medical Research Council (mMRC) dyspnoea scale | 8 weeks and 12weeks
  The mMRC scale is a five-category scale to characterize the level of dyspnoea with physical activity in which higher scores correspond with increased dyspnoea.
The change of EuroQol five-dimension five-level (EQ-5D-5L)5L) questionnaire and it's Visual Analogue Scale (VAS) | 8 weeks and 12weeks
  To evaluate patients quality of life (QoL) by using EQ-5D-5L, higher score better QoL. EuroQol Visual Analogue Scale assess generic health ranging from 0-100, higher score better health experience.
Pulmonary function assessment on FEV1, FVC, and FEV1/FVC ratio | 8 weeks
  FEV1, FVC, and FEV1/FVC ratio will be measured with the Air Next Spirometer (NuvoAir, Sweden) in combination with the mobile coaching system. The higher of FEV1/FVC ratio, the healthier of subjects.
Adverse event assessment | 8 weeks and 12weeks
  Any reported adverse event related to study treatment will be analyzed throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiu Lin, PhD, Principal Investigator — Hong Kong Institute of Integrative Medicine
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

REFERENCES:
- [Derived] Sum CH, Ching JYL, Song T, Cheong PK, Lo CW, Lai MK, Chia CP, Chan KL, Mak WY, Leung KC, Leung SB, Zhang H, Lin Z. Chinese medicine for residual symptoms of COVID-19 recovered patients (long COVID)-A double-blind, randomized, and placebo-controlled clinical trial protocol. Front Med (Lausanne). 2023 Jan 4;9:990639. doi: 10.3389/fmed.2022.990639. eCollection 2022. PMID 36687403